CLINICAL TRIAL: NCT01952093
Title: Effects of Early Intervention for Preterm Children at School Age
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 201112106RIB
Record Dates: First submitted 2013-09-18; First posted 2013-09-27 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2016-04

CONDITIONS: Premature Birth
Keywords: Early intervention; Mother-child interaction; Neurodevelopment; Parenting; Prematurity; School age
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Usual care program: VLBW preterm infants who received usual medical care during hospitalization after birth.(in the previous study)
- Clinic-based intervention program: VLBW preterm infants who received specific early intervention program delivered at clinic before 1 year of corrected age (in the previous study)
  Interventions: Behavioral: Clinic-based intervention program
- Home-based intervention program: VLBW preterm infants who received specific early intervention program delivered at home before 1 year of corrected age (in the previous study)
  Interventions: Behavioral: Home-based intervention program
- Term control group: Healthy term infants

INTERVENTIONS:
Behavioral: Home-based intervention program — The intervention had been done in the previous intervention study. The intervention included in-hospital and after-discharge service. After-discharge intervention performed at 0, 1, 2, 4, 6, 9, 12 months of age at the home.
  Other Names: HBIP
  Groups: Home-based intervention program
Behavioral: Clinic-based intervention program — The intervention had been done in the previous intervention study. The intervention included in-hospital and after-discharge service. After-discharge intervention performed at 0, 1, 2, 4, 6, 9, 12 months of age at the clinic.
  Other Names: CBIP
  Groups: Clinic-based intervention program

SUMMARY:
Despite the remarkable achievements in neonatal survival of preterm infants with very low birth weight (VLBW, birth weight < 1,500 g) over the past three decades, improvements have produced little change in their prevalence of severe developmental disability and the rate of low severity dysfunctions (e.g., learning disabilities, low IQ, attention-deficit hyperactivity disorder, specific neuropsychological deficits, poor perceptual-motor skills and internalizing behavioral problems) remains high as 50% to 70%. Few intervention programs developed for preterm infants in Western societies were shown to have short- to long-term benefits in certain cognitive functions, however, rare studies have investigated intervention effect at school age and explored plausible neurological pathway for effective intervention. This three-year study was therefore aimed to extend our previous research to longitudinally examine the effectiveness of three intervention programs (clinic-based intervention program [CBIP], home-based intervention program [HBIP] and usual care program [UCP]) for VLBW preterm children in Taiwan at seven years of age.(The intervention had been delivered from birth to one year of corrected age in the previous study. The intervention will not be given in this study.)The CBIP and HBIP contained similar child- and parent-focused services as well as interaction activities but were respectively delivered at the clinic for the CBIP and at home for the HBIP. A total of 178 VLBW preterm infants had been randomly assigned to the CBIP, HBIP or UCP. Sixty-two gender and maternal education level matched term children with normal birth weight had also been included to serve as the reference group for comparison of developmental outcomes. Effectiveness examined included child and parent outcomes. The long-term effect of the early intervention for preterm children would provide important information to help medical professionals and public policy makers to develop an effective intervention for Taiwanese preterm children who are at risk of developmental disorders.

DETAILED DESCRIPTION:
Specific Aims:

This study was to extend our previous research to longitudinally examine the effectiveness of three intervention programs (CBIP, HBIP and UCP) for VLBW preterm children in Taiwan at seven years of age. Gender and maternal education level matched term children were also included to serve as the reference group for comparison of developmental outcomes. The intervention had been delivered from birth to one year of corrected age in the previous study. Effectiveness examined including children's and parental outcomes. Primary outcome referred to measures of child neurobehavioral functions. Neurobehavioral assessment included cognitive, motor and behavioral measurement. Secondary outcomes referred to child growth and health, neurophysiological functions, and the quality of parenting measures. Neurophysiological assessment referred to electroencephalogram/event-related potential examinations that were used to investigate the neurological pathways underlying the effective intervention.

Subjects and Methods:

Participants:

One hundred and seventy-eight VLBW preterm children and 62 term children who had participated in our previous study were enrolled in this study. VLBW preterm children were born or admitted at the National Taiwan University Hospital, the Mackay Memorial Hospital and Taipei City Hospital, Branch for Women and Children in Taipei, Taiwan, during the time period of 2006 to 2008.

Methods:

While age seven is an important time period that children enter elementary school and begin to participate in school activities, more comprehensive outcome measurements are required. The World Health Organization emphasizes that health conditions should be considered from the body, individuals and societal perspectives as depicted in the International Classification of Functioning, Disability and Health model. Accordingly, the outcome measures in this study consisted of the primary (i.e., child neurobehavioral functions) and secondary outcomes (i.e., child growth and health, neurophysiological functions, and quality of parenting). Child neurobehavioral assessment included measurements of cognitive, motor, and behavior function. The domains of cognitive functions examined including the intelligence (IQ test), the efficiency of attention control (sustained attention test), and the cognitive flexibility and planning (executive function test). The motor function included motor skill acquisition and coordination. Children's behavior was measured using the parental report of child behavior and teacher's observation for child's adaptive behavior in the school context. Children's educational resources (special education or resource class) or other education-related support received from any institution would also be recorded in this study. Child neurophysiological functions were measured by the electroencephalogram (EEG)/event-related potential (ERP) technique.

All families were contacted via phone call and mail to be enrolled in this study. Children and their parents would have been examined for the following outcomes when the children approached at seven years of age. All measures except for the neurophysiological measures were conducted at Infant Motor Development Laboratory, School of Physical Therapy, National Taiwan University. Several examiners with the background knowledge of physical therapy or psychology received training with the testing instruments and procedures. Before commencing the study assessments, the interrater reliability (agreement with an experienced investigator > 0.80) would have been required for the assessors. All the examiners were kept blind to children's group assignment. To decrease the fatigue in children due to the prolonged examination, participants were asked to return twice for assessment.The first assessment would have taken 180 minutes which consisted of the IQ test, sustained attention test, and executive function test that the whole session.The second assessment was the neurophysiological measurement with the EEG/ERP tasks which would have taken 90 minutes.

ELIGIBILITY:
Seven years old children who received the intervention service in our previous intervention study will be invited to participate in this study.

* The inclusion criteria for term infants were: birth weight greater than 2500 g, gestational age within 38-42 weeks, and the absence of serious prenatal and perinatal complications.
* The inclusion criteria for VLBW preterm infants were: birth weight less than 1500 g, gestational age less than 37 weeks, and the singleton or the first child of twin/multiple birth.
* The exclusion criteria for VLBW preterm infants were: admission to the study hospitals >7 days of birth and infants with congenital anomalies or severe neonatal diseases.
* Infants exhibiting persistently unstable physiological conditions until 36 weeks' post- menstrual age (PMA) or older, being discharged from hospital at 44 weeks' PMA or older, or developing severe neonatal diseases (e.g., seizure, hydrocephalus, ventriculoperitoneal shunt, periventricular leukomalacia, grade III-IV intraventricular hemorrhage, necrotizing enterocolitis with colostomy, and stage IV-V retinopathy of prematurity) were early terminated in this study.
* Additional selection criteria for all infants in this study were as follows: mothers who read and speak Chinese, maternal age older than 18 years, absence of maternal alcohol or drug abuse history, and parents married at child's birth.

Ages: 7 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Term and VLBW preterm children were born at the National Taiwan University Hospital and the Mackay Memorial Hospital (MMH) and who received the intervention service in our previous intervention study will be invited to participate in this study.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Child neurobehavioral development | at 7 years of age
  Child neurobehavioral assessment including cognitive and, motor, and behavior functions.
  Cognitive functions were assessed by the intelligence (IQ test), the efficiency of attention control (sustained attention test), and the cognitive flexibility and planning (executive function test).
  Motor functions assessment included motor skill acquisition and coordination. Child's behavior was measured by the parent/teacher reported questionnaire (two different versions) of child's adaptive behavior in the school context.

SECONDARY OUTCOMES:
Parenting | at 7 years of age
  The parental outcome was measured with the quality of parenting.
Child health condition | at 7 years of age
  Child health condition were measured by a parent report questionnaire and chart review.
Child neurophysiological functions | at 7 years of age
  Child's neurophysiological functions were measured by the electroencephalogram (EEG)/event-related potential (ERP) technique for the participating children.
Child educational resources | at 7 years of age
  The utility of special education and resource classes and the receiving of other educational support from any institution were also be recorded in this study.
Child growth-weight | at 7 years of age
  Child's weight was measured by electronic weighting scale in kilogram
Child growth-height | at 7 years of age
  Child's weight was measured by Kidmeasure in centimeter

CONTACTS AND LOCATIONS:
Overall Officials: Suh-Fang Jeng, Sc.D, Principal Investigator — School of Physical Therapy, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No